CLINICAL TRIAL: NCT03590600
Title: A Randomized, Double Blind, Placebo-controlled, Single Ascending Dose Study to Evaluate Safety, Tolerability, and Pharmacokinetics of Single Doses of BTZ043 in Healthy Adult Volunteers
Brief Title: A Single Ascending Dose Study of BTZ043
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Michael Hoelscher (Other)
Collaborators: German Center for Infection Research (Other); German Federal Ministry of Education and Research (Other Government); Hans Knöll Institute (HKI) (Unknown)
Responsible Party: Sponsor-Investigator, Michael Hoelscher, Director, Ludwig-Maximilians - University of Munich
Organization: Ludwig-Maximilians - University of Munich (Other)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LMU-IMPH-BTZ043-01
Record Dates: First submitted 2018-06-04; First posted 2018-07-18 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Tuberculosis; Tuberculosis, Pulmonary; Bacterial Infections; Lung Diseases; Mycobacterium Infections
Keywords: Phase 1; Anti-Bacterial Agents; Respiratory Tract Infections
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Pulmonary; Bacterial Infections; Lung Diseases; Mycobacterium Infections; Respiratory Tract Infections | interventions — 2-(2-methyl-1,4-dioxa-8-azaspiro(4.5)dec-8-yl)-8-nitro-6-(trifluoromethyl)-4H-1,3-benzothiazin-4-one

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Subjects, investigators and investigators' staff, persons performing the assessments or being responsible for determining dosing regimen/adjustments, and staff of the sponsor or data analysts, will remain blinded from the time of randomization until database lock, using the following methods: randomization data, including any documentation identifying the treatment allocation, are kept strictly confidential until the time of unblinding with the following exceptions: staff responsible for study drug management (i.e. the staff in the CRO CTS department preparing the IMP).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Cohort 1: 125 mg BTZ-043 fasting (Experimental): N=8, 125 mg BTZ-043 fasting, oral administration, powder and solvent for oral suspension, single dose
  Interventions: Drug: BTZ-043
- Cohort 1: Placebo (Placebo Comparator): N=2, matching placebo, powder and solvent for oral solution, single dose
  Interventions: Drug: Placebo
- Cohort 2: 250 mg BTZ-043 fasting (Experimental): N=8, 250 mg BTZ-043 fasting, oral administration, powder and solvent for oral suspension, single dose
  Interventions: Drug: BTZ-043
- Cohort 2: Placebo (Placebo Comparator): N=2, matching placebo, powder and solvent for oral solution, single dose
  Interventions: Drug: Placebo
- Cohort 3: 500 mg BTZ-043 fasting (Experimental): N=8, 500 mg BTZ-043 fasting, oral administration, powder and solvent for oral suspension, single dose
  Interventions: Drug: BTZ-043
- Cohort 3: Placebo (Placebo Comparator): N=2, matching placebo, powder and solvent for oral solution, single dose
  Interventions: Drug: Placebo
- Cohort 4: 1000 mg BTZ-043 fasting (Experimental): N=8, 1000 mg BTZ-043 fasting, oral administration, powder and solvent for oral suspension, single dose
  Interventions: Drug: BTZ-043
- Cohort 4: Placebo (Placebo Comparator): N=2, matching placebo, powder and solvent for oral solution, single dose
  Interventions: Drug: Placebo
- Cohort 5: 2000mg BTZ-043 fasting (Experimental): N=8, 2000 mg BTZ-043 fasting, oral administration, powder and solvent for oral suspension, single dose
  Interventions: Drug: BTZ-043
- Cohort 5: Placebo (Placebo Comparator): N=2, matching placebo, powder and solvent for oral solution, single dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BTZ-043 — Powder and solvent for oral suspension
  Arms: Cohort 1: 125 mg BTZ-043 fasting; Cohort 2: 250 mg BTZ-043 fasting; Cohort 3: 500 mg BTZ-043 fasting; Cohort 4: 1000 mg BTZ-043 fasting; Cohort 5: 2000mg BTZ-043 fasting
Drug: Placebo — Matching placebo: powder and solvent for oral suspension
  Arms: Cohort 1: Placebo; Cohort 2: Placebo; Cohort 3: Placebo; Cohort 4: Placebo; Cohort 5: Placebo

SUMMARY:
This study is a randomized, double-blind, placebo-controlled, single ascending dose study to evaluate safety, tolerability, and pharmacokinetics of single doses of BTZ043 in healthy adult volunteers. The study is conducted at a study centre in Germany. Up to 50 male and female participants will be included in this study in up to 5 cohorts; each cohort will consist of 10 subjects: in each cohort 8 subjects will be assigned to BTZ-043 and 2 to placebo. The doses tested will be: 125mg, 250mg, 500mg, 1000mg and 2000mg. Safety will be assessed via regular vital sign measurement, 12-lead ECG parameters, physical examination and safety laboratory assessments.

Subjects will be hospitalized from Day -1 until discharge in the morning of Day 3. After completion of all Day 3 assessments of a cohort, blinded safety data will be reviewed and the next dose increment will be decided by the Trial Steering Committee (TSC).

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent
* Healthy male or female subjects aged between ≥18 and ≤55 years at screening who are able to read, write, and fully understand the German language
* BMI between ≥18 and ≤30 kg/m2, with a body weight between ≥55 and ≤90 kg at screening
* Vital signs within range: pulse rate 50-90 bpm, systolic blood pressure 90-140 mmHg, diastolic blood pressure 50-90 mmHg
* No clinically significant findings in laboratory tests
* Women must be of non-childbearing potential, that is, either postmenopausal or premenopausal with documented tubal ligation or hysterectomy or women who are at least 6 weeks post-surgical bilateral oophorectomy
* Male subjects must agree to use a condom with spermicide when engaging in sexual intercourse during the study period and for 2 months after study drug dosing, if they have not had a vasectomy at least 6 months before study start
* Male subjects must not donate sperm during the study and for 2 months after study drug dosing
* Able to swallow the amount of drug in succession
* Agree not to donate blood (or bloodcomponents) until 1 month after receiving study drug
* Normal consumption of alcohol
* Willing to forgo sunbathing and prolonged exposure to sunlight during the study period
* Willing to forgo strenuous exercise from 72 hours prior to admission until discharge

Exclusion Criteria:

* Any known chronic systemic viral infection
* Any relevant systemic infection or other systemic illness
* Vaccination 30 days prior to drug administration
* Known hypersensitivity to any of the excipients of the study drug
* A clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, hematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, endocrine, connective tissue diseases or disorders, or have a clinically relevant surgical history or any other medical condition
* History of or current alcohol or illicit drug abuse
* Positive results in the urine drug screen or blood alcohol test at admission
* Current or recent (within the past 3 months before drug administration) use of tobacco or other nicotine-containing product or positive results of cotinine test at screening or admission
* Use of any prescription or over-the-counter (OTC) drug or herbal product within 14 days before drug administration with exception for sporadic use of ibuprofen or paracetamol for example in case of pain
* Use of any known drug metabolism enzyme-altering drug or supplement within 14 days before dosing or consumption of foods or beverages containing grapefruit within 48 hours before admission
* ECG findings in the screening ECG of QTcF-interval over 450 ms; atrioventricular (AV) block with PR-interval over 200 ms, prolongation of the QRS complex over 120 ms, or other changes in the ECG that are clinically relevant as per discretion of the investigator
* Long QT syndrome, or family history of long QT syndrome or sudden death of unknown or cardiac-related cause
* Use or planned necessary use of any QT-prolonging agents
* Participation in another investigational drug study within the previous 30 days before drug administration
* Any donation of blood, plasma, or platelets or significant loss of blood within the previous 30 days before drug administration
* Previous randomization in this study
* Volunteer unwilling or unable to comply with protocol requirements in the judgment of the investigator
* Vulnerable subject (e.g. person is kept in detention)
* Employees of the sponsor or subjects who are employees or relatives of the investigator

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-06-07 (Actual); Primary Completion 2018-08-14 (Actual); Study Completion 2019-03-05 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events concerning ECG as assessed by CTCAE v4.03 (Common Terminology Criteria for Adverse Events) | 0.5 hours to 12.0 hours post-dosing
  Measured by 12-lead ECG assessments on 6 different timepoints.
Number of participants with treatment-related adverse events concerning safety laboratory as assessed by CTCAE v4.03 | 24 hours to 26 hours post-dosing
  Measured by clinical chemistry, haematology, coagulation, urinalysis on 2 different timepoints
Number of participants with treatment-related adverse events concerning vital signs as assessed by CTCAE v4.03 | 0.25 hours to 48 hours post-dosing
  Measured by blood pressure, pulse rate, respiratory rate and tympanic body temperature on 7 different timepoints
Number of participants with treatment-related adverse events concerning clinical observations as assessed by CTCAE v4.03 | 4 hours to 48 hours post-dosing
  Examination of general appearance, skin, neck (including thyroid), throat, lungs, heart, abdomen, back, lymph nodes, extremities, vascular and neurological systems.

SECONDARY OUTCOMES:
Pharmacokinetic assessment of BTZ-043 after a single oral dose | 0.25 hours to 36 hours post-dosing
  Blood samples for the determination of Area under the plasma concentration versus time curve (AUC) will be assessed in BTZ-043 and the metabolites BTZ-045S and M2
Pharmacokinetic assessment of BTZ-043 after a single oral dose | 0.25 hours to 36 hours post-dosing
  Blood samples for the determination of Peak Plasma Concentration (Cmax) will be assessed in BTZ-043 and the metabolites BTZ-045S and M2
Determining the effect of sex differences on systemic exposure by analyzing the PK of BTZ-043 in male and female participants. | 0.25 hours to 36 hours post-dosing
  Estimated via comparison of the exposure (AUC0-inf) of BTZ-043 in males and females

CONTACTS AND LOCATIONS:
Locations (1):
- Nuvisan, Neu-Ulm, Bavaria, Germany